CLINICAL TRIAL: NCT02030535
Title: A Randomised, Placebo-controlled, Double-blind, Single Dose, Cross-over Study to Evaluate the Efficacy and Safety of Orally Inhaled Tiotropium + Olodaterol as Both a Fixed Dose Combination and a Free Combination (Both Delivered by the Respimat® Inhaler) in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Study to Evaluate the Effect on Lung Function and ECG When a Combination of Tiotropium Plus Olodaterol is Administered to Patients With COPD Either From a Single Inhaler or Each Compound is Administered After Each Other From Two Different Inhalers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1237.7; 2013-002652-32 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-01-07; First posted 2014-01-08 (Estimated); Results first posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol; Tiotropium Bromide

ARMS (3):
- Tiotropium/Olodaterol FDC (Experimental): patient will receive tiotropium and olodaterol in a fixed dose combination
  Interventions: Drug: tiotropium; Drug: olodaterol
- Tiotropium and Olodaterol FC (Experimental): patient will receive tiotropium and olodaterol in a free combination
  Interventions: Drug: olodaterol; Drug: tiotropium
- Placebo (Placebo Comparator): patient will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: olodaterol — free combination with tiotropium
  Arms: Tiotropium and Olodaterol FC
Drug: tiotropium — free combination with olodaterol
  Arms: Tiotropium and Olodaterol FC
Drug: Placebo
  Arms: Placebo
Drug: tiotropium — fixed dose combination with olodaterol
  Arms: Tiotropium/Olodaterol FDC
Drug: olodaterol — fixed dose combination with tiotropium
  Arms: Tiotropium/Olodaterol FDC

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of orally inhaled tiotropium and olodaterol as both a fixed dose combination and a free combination with respect to lung function and ECG parameters

ELIGIBILITY:
Inclusion criteria:

* patients must sign informed consent consistent with ICH-GCP guidelines prior to participation in the trial, which includes medication washout and restrictions.
* Patients must have a diagnosis of COPD and must meet the following spirometric criteria:

Patients must have relatively stable airway obstruction with a post-bronchodilator (10 to 45 minutes after 400mcg salbutamol) FEV1>30% and < 80% of predicted normal (ECSC, GOLD II - III) and a post-bronchodilator FEV1/FVC <70% at Visit 1

* Male or female patients, 40 years of age or older.
* Patients must be current or ex-smokers with a smoking history of more than 10 pack years.
* Patients who have never smoked cigarettes must be excluded.
* Patients must be able to perform technically acceptable pulmonary function tests according to ATS/ERS guidelines and maintain records in a paper diary
* Patients must be able to inhale medication in a competent manner from the RESPIMAT inhaler and from a metered dose inhaler (MDI).

Exclusion criteria:

* Significant disease other than COPD
* Clinically relevant abnormal lab values.
* History of asthma.
* Diagnosis of thyrotoxicosis
* Diagnosis of paroxysmal tachycardia
* History of myocardial infarction within 1 year of screening visit
* Unstable or life-threatening cardiac arrhythmia
* Hospitalization for heart failure within the past year
* Known active tuberculosis
* Malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years
* History of life-threatening pulmonary obstruction and patients with chronic respiratory failure
* History of cystic fibrosis
* Clinically evident bronchiectasis
* History of significant alcohol or drug abuse
* Thoracotomy with pulmonary resection
* Patients treated with oral or patch ß-adrenergics
* Patients treated with oral corticosteroid medication at unstable doses or at doses in excess of 10mg prednisolone per day or equivalent
* Regular use of daytime oxygen therapy for more than one hour per day
* Pulmonary rehabilitation program in the six weeks prior to the screening visit or patients currently in a pulmonary rehabilitation program
* Investigational drug within one month or six half lives (whichever is greater) prior to screening visit
* Known hypersensitivity to ß-adrenergic and/or anticholinergic drugs, BAC, EDTA
* Pregnant or nursing women
* Women of childbearing potential not using a highly effective method of birth control
* Patient who have previously been randomized in this study or are currently participating in another study
* Patients who are unable to comply with pulmonary medication restrictions prior to randomization

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (6):
- Germany (6):
  - 1237.7.49004 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.7.49005 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.7.49007 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1237.7.49002 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 1237.7.49003 Boehringer Ingelheim Investigational Site, Hamburg
  - 1237.7.49001 Boehringer Ingelheim Investigational Site, Weinheim

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: Total number of patients randomised and treated in the study. (This is a cross-over trial consisting of a minimum two-week screening period. After screening, eligible patients were randomly assigned to one of 12 treatment sequences. Each patient received all three treatments as single doses on the three test days. Between test days with single dose administration there are 3-week washout periods.)
Period: Treatment Period 1 (1 Day)
Arm/Group | Overall Study
Started | 53
Completed | 53
Not Completed | 0
Period: Washout Period 1 (21 Days)
Arm/Group | Overall Study
Started | 53
Completed | 52
Not Completed | 1
Not completed — Adverse Event | 1
Period: Treatment Period 2 (1 Day)
Arm/Group | Overall Study
Started | 52
Completed | 52
Not Completed | 0
Period: Washout Period 2 (21 Days)
Arm/Group | Overall Study
Started | 52
Completed | 52
Not Completed | 0
Period: Treatment Period 3 (1 Day)
Arm/Group | Overall Study
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This patient set included all randomised patients who were administered study medication.
Groups:
- Overall Study: Total number of patients randomised and treated in the study.
Arm/Group | Overall Study
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 31

OUTCOME MEASURES:

1. Secondary Outcome: Mean (Heart Rate Corrected QT Interval (Using Fredericia Adjustment)) QTcF Interval Change From Patient Baseline Over All Post-dose Time Points
Description: Mean QTcF interval change from patient baseline over all post-dose time points (5min, 10min, 25min and 50min)
Time Frame: 40 min pre-dose and at 5 min, 10 min, 25 min and 50 min post-dose
Population: Treated set (observed cases)
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Placebo: Single test dose of oral inhalation of Placebo via RESPIMAT inhaler.
  2 inhalations a.m. dosing.
- Tio+Olo 5/5μg: Single test dose of oral inhalation of Tio+Olo FDC(fixed dose combination) (5/5 μg) inhalation solution as fixed dose inhalation solution (Tio+Olo FDC) 2.5 μg each per actuation.
  2 inhalations a.m. dosing via RESPIMAT® inhaler
- Tiotropium 5μg + Olodaterol 5μg: Single test dose of oral inhalation of tiotropium (5 μg) and olodaterol (5 μg) free combination (FC) (Tio/Olo free combination)
  Olodaterol: 5 μg (2.5 μg per actuation)
  Tiotropium: 5 μg (2.5 μg per actuation)
  2 inhalations a.m. dosing via RESPIMAT® inhaler
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 52 | 52 | 52
ms | 1.3 (7.1) | 2.2 (6.9) | 1.9 (6.9)

2. Secondary Outcome: Peak QTcF Interval Change From Patient Baseline Over All Post-dose Time Points
Description: Peak QTcF interval change from patient baseline over all post-dose time points (5min, 10min, 25min and 50min)
Time Frame: 40 min pre-dose and at 5 min, 10 min, 25 min and 50 min post-dose
Population: Treated set (observed cases)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 52 | 52 | 52
ms | 5.2 (8.3) | 5.7 (7.6) | 5.7 (7.3)

3. Secondary Outcome: Mean Heart Rate Change From Patient Baseline Over All Post-dose Time Points
Description: Mean heart rate change from patient baseline over all post-dose time points (5min, 10min, 25min and 50min)
Time Frame: 40 min pre-dose and at 5 min, 10 min, 25 min and 50 min post-dose
Population: Treated set (observed cases)
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 52 | 52 | 52
bpm | -3.0 (5.2) | -2.5 (5.5) | -3.6 (4.3)

4. Secondary Outcome: Peak Heart Rate Change From Patient Baseline Over All Post-dose Time Points
Description: Peak heart rate change from patient baseline over all post-dose time points (5min, 10min, 25min and 50min)
Time Frame: 40 min pre-dose and at 5 min, 10 min, 25 min and 50 min post-dose
Population: Treated set (observed cases)
Measure: Mean (Standard Deviation); unit: bpm
Groups:
- Tio+Olo 5/5μg: Single test dose of oral inhalation of Tio+Olo FDC(fixed dose combination) (5/5 μg) inhalation solution as fixed dose inhalation solution (Tio+Olo FDC) 2.5 μg each per actuation.
  2 inhalations (a.m. dosing) via RESPIMAT® inhaler
- Tiotropium 5μg + Olodaterol 5μg: Single test dose of oral inhalation of tiotropium (5 μg) and olodaterol (5 μg) free combination (FC) (Tio/Olo free combination)
  Olodaterol: 5 μg (2.5 μg per actuation)
  Tiotropium: 5 μg (2.5 μg per actuation)
  2 inhalations (a.m. dosing) via RESPIMAT® inhaler
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 52 | 52 | 52
bpm | -0.7 (5.5) | -0.3 (5.7) | -1.2 (4.4)

5. Primary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under the Curve (AUC) (0-3hours) Response After Single-dose Administration
Description: The response was defined as the change from patient baseline. Patient baseline was the average of the mean pre-dose values (period baseline) on each test day (Visit 2 (Day 1), Visit 3 (Day 22 (±7days)), and Visit 4 (Day 43±7days)).
  For patients who did not complete all periods, patient baseline was the average of the available period baselines.
  The means presented are the adjusted means.
Time Frame: 1 hour (h) and 10 min pre-dose and at 15 min, 30 min, 1 h, 2 h and 3 h post-dose
Population: Full Analysis Set (FAS): This patient set included all patients in the TS who had at least 1 visit (Visit 2(Day1), Visit 3(Day22), or Visit 4(Day43)) with both the period baseline value plus any evaluable post-dose spirometry measurement from the same visit.
Measure: Mean (Standard Error); unit: Litres
Groups:
- Placebo: Single test dose of oral inhalation of Placebo via RESPIMAT inhaler.
  2 inhalations ante meridiem (a.m.) dosing.
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 53 | 52 | 52
Litres | 0.014 (0.016) | 0.233 (0.016) | 0.266 (0.016)
Statistical Analysis 1: Comparison: Placebo vs Tio+Olo 5/5μg; Test type: Superiority or Other; p < 0.0001, Mixed models repeated measures analysis — Mixed effect model repeated measures (MMRM) including fixed effects of treatment and period; patient baseline and period baseline as covariates; patient as a random effect; Kenward-Roger approximation of denominator degrees of freedom. Compound symmetry covariance structure for within-patient variation; Adjusted mean difference = 0.219, 95% CI 2-sided [0.187 to 0.252], Standard Error of Mean 0.016 — Tio+Olo 5/5μg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Tiotropium 5μg + Olodaterol 5μg; Test type: Superiority or Other; p < 0.0001, Mixed models repeated measures analysis — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 5, analysis 1]; Adjusted mean difference = 0.252, 95% CI 2-sided [0.220 to 0.284], Standard Error of Mean 0.016 — Tiotropium 5μg + Olodaterol 5μg minus Placebo
Statistical Analysis 3: Comparison: Tio+Olo 5/5μg vs Tiotropium 5μg + Olodaterol 5μg; Descriptive comparison. Statistical Analyses 1 & 2 were included in the hierarchical testing sequence (alpha protected), and analysis 3 was not included in the hierarchical testing sequence (not alpha protected); Test type: Superiority or Other; Adjusted mean difference = -0.033, 95% CI 2-sided [-0.065 to -0.001], Standard Error of Mean 0.016 — Tio+Olo 5/5μg minus Tiotropium 5μg + Olodaterol 5μg

6. Secondary Outcome: Heart Rate Change From Patient Baseline at Individual Post-dose Time Points
Description: Heart rate change from patient baseline at individual post-dose time points
Time Frame: 40 min pre-dose and at 5 min, 10 min, 25 min and 50 min post-dose
Population: Treated set (observed cases)
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 52 | 52 | 52
bpm
  5 min | -2.3 (5.2) | -2.5 (5.5) | -2.9 (4.6)
  10 min | -2.7 (5.9) | -2.4 (5.5) | -3.1 (4.6)
  25 min | -3.1 (5.5) | -2.6 (6.0) | -4.5 (5.0)
  50 min | -4.1 (5.6) | -2.4 (6.0) | -3.9 (4.7)

7. Secondary Outcome: Mean RR (Time Interval of ECG) Change From Patient Baseline Over All Post-dose Time Points
Description: Mean RR change from patient baseline over all post-dose time points (5min, 10min, 25min and 50min)
Time Frame: 40 min pre-dose and at 5 min, 10 min, 25 min and 50 min post-dose
Population: Treated set (observed cases)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 52 | 52 | 52
ms | 40.4 (57.7) | 29.3 (57.1) | 39.5 (51.5)

8. Secondary Outcome: Peak RR Change From Patient Baseline Over All Post-dose Time Points
Description: Peak RR change from patient baseline over all post-dose time points (5min, 10min, 25min and 50min)
Time Frame: 40 min pre-dose and at 5 min, 10 min, 25 min and 50 min post-dose
Population: Treated set (observed cases)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 52 | 52 | 52
ms | 68.8 (64.3) | 55.5 (59.5) | 68.0 (52.7)

9. Secondary Outcome: RR Change From Patient Baseline at Individual Post-dose Time Points
Description: RR change from patient baseline at individual post-dose time points
Time Frame: 40 min pre-dose and at 5 min, 10 min, 25 min and 50 min post-dose
Population: Treated set (observed cases)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 52 | 52 | 52
ms
  5 min | 29.9 (62.5) | 29.7 (58.5) | 31.9 (55.5)
  10 min | 38.8 (68.9) | 28.1 (57.4) | 33.5 (56.1)
  25 min | 40.4 (59.4) | 33.0 (65.7) | 50.0 (59.9)
  50 min | 52.3 (62.7) | 25.2 (64.9) | 44.0 (57.0)

10. Secondary Outcome: Mean QT (Time Interval of ECG) Change From Patient Baseline Over All Post-dose Time Points
Description: Mean QT change from patient baseline over all post-dose time points (5min, 10min, 25min and 50min)
Time Frame: 40 min pre-dose and at 5 min, 10 min, 25 min and 50 min post-dose
Population: Treated set (observed cases)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 52 | 52 | 52
ms | 7.2 (10.7) | 6.5 (11.1) | 7.9 (9.9)

11. Secondary Outcome: Peak QT (Time Interval of ECG) Change From Patient Baseline Over All Post-dose Time Points
Description: Peak QT change from patient baseline over all post-dose time points (5min, 10min, 25min and 50min)
Time Frame: 40 min pre-dose and at 5 min, 10 min, 25 min and 50 min post-dose
Population: Treated set (observed cases)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 52 | 52 | 52
ms | 12.4 (11.5) | 11.5 (11.1) | 13.4 (10.6)

12. Secondary Outcome: QT Change From Patient Baseline at Individual Post-dose Time Points
Description: QT change from patient baseline at individual post-dose time points
Time Frame: 40 min pre-dose and at 5 min, 10 min, 25 min and 50 min post-dose
Population: Treated set (observed cases)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 52 | 52 | 52
ms
  5 min | 4.3 (10.7) | 5.5 (11.2) | 4.9 (10.4)
  10 min | 7.1 (12.6) | 6.3 (11.8) | 7.9 (11.3)
  25 min | 7.9 (11.4) | 7.4 (12.0) | 9.6 (11.1)
  50 min | 9.4 (12.1) | 6.7 (12.6) | 9.4 (10.9)

13. Secondary Outcome: Mean QTcB (Heart Rate Corrected QT Interval (Using Bazett Adjustment)) Change From Patient Baseline Over All Post-dose Time Points
Description: Mean QTcB (Heart Rate Corrected QT Interval (Using Bazett Adjustment))change from patient baseline over all post-dose time points (5min, 10min, 25min and 50min)
Time Frame: 40 min pre-dose and at 5 min, 10 min, 25 min and 50 min post-dose
Population: Treated set (observed cases)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 52 | 52 | 52
ms | -1.9 (9.0) | -0.2 (8.6) | -1.4 (8.1)

14. Secondary Outcome: Peak QTcB (Heart Rate Corrected QT Interval (Using Bazett Adjustment)) Change From Patient Baseline Over All Post-dose Time Points
Description: Peak QTcB (Heart Rate Corrected QT Interval (Using Bazett Adjustment))change from patient baseline over all post-dose time points (5min, 10min, 25min and 50min)
Time Frame: 40 min pre-dose and at 5 min, 10 min, 25 min and 50 min post-dose
Population: Treated set (observed cases)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 52 | 52 | 52
ms | 3.0 (10.7) | 4.2 (9.7) | 3.5 (8.5)

15. Secondary Outcome: QTcB Change From Patient Baseline at Individual Post-dose Time Points
Description: QTcB change from patient baseline at individual post-dose time points
Time Frame: 40 min pre-dose and at 5 min, 10 min, 25 min and 50 min post-dose
Population: Treated set (observed cases)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 52 | 52 | 52
ms
  5 min | -2.5 (9.0) | -1.4 (8.8) | -2.6 (8.7)
  10 min | -1.4 (9.9) | -0.2 (8.7) | -0.0 (9.0)
  25 min | -1.0 (11.3) | 0.1 (10.3) | -2.2 (9.3)
  50 min | -2.6 (9.9) | 0.7 (9.8) | -0.7 (9.4)

16. Secondary Outcome: Mean PR (Time Interval of ECG) Change From Patient Baseline Over All Post-dose Time Points
Description: Mean PR change from patient baseline over all post-dose time points (5min, 10min, 25min and 50min)
Time Frame: 40 min pre-dose and at 5 min, 10 min, 25 min and 50 min post-dose
Population: Treated set (observed cases)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 52 | 52 | 52
ms | 0.6 (4.9) | 1.6 (6.3) | 1.4 (6.4)

17. Secondary Outcome: Peak PR (Time Interval of ECG) Change From Patient Baseline Over All Post-dose Time Points
Description: Peak PR change from patient baseline over all post-dose time points (5min, 10min, 25min and 50min)
Time Frame: 40 min pre-dose and at 5 min, 10 min, 25 min and 50 min post-dose
Population: Treated set (observed cases)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 52 | 52 | 52
ms | 3.9 (4.8) | 4.6 (5.9) | 4.7 (7.2)

18. Secondary Outcome: PR Change From Patient Baseline at Individual Post-dose Time Points
Description: PR change from patient baseline at individual post-dose time points
Time Frame: 40 min pre-dose and at 5 min, 10 min, 25 min and 50 min post-dose
Population: Treated set (observed cases)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 52 | 52 | 52
ms
  5 min | 0.1 (5.9) | 1.2 (7.3) | -0.2 (6.6)
  10 min | 0.1 (6.0) | 2.5 (8.4) | 1.4 (7.1)
  25 min | 0.1 (6.5) | 0.8 (6.3) | 1.9 (7.8)
  50 min | 2.2 (5.4) | 1.9 (5.4) | 2.7 (7.7)

19. Secondary Outcome: Mean QRS (Time Interval of ECG) Change From Patient Baseline Over All Post-dose Time Points
Description: Mean QRS change from patient baseline over all post-dose time points (5min, 10min, 25min and 50min)
Time Frame: 40 min pre-dose and at 5 min, 10 min, 25 min and 50 min post-dose
Population: Treated set (observed cases)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 52 | 52 | 52
ms | -0.3 (1.3) | 0.1 (1.5) | 0.1 (1.3)

20. Secondary Outcome: Peak QRS (Time Interval of ECG) Change From Patient Baseline Over All Post-dose Time Points
Description: Peak QRS change from patient baseline over all post-dose time points (5min, 10min, 25min and 50min)
Time Frame: 40 min pre-dose and at 5 min, 10 min, 25 min and 50 min post-dose
Population: Treated set (observed cases)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 52 | 52 | 52
ms | 0.6 (1.5) | 0.9 (1.5) | 1.0 (1.3)

21. Secondary Outcome: QRS Change From Patient Baseline at Individual Post-dose Time Points
Description: QRS change from patient baseline at individual post-dose time points
Time Frame: 40 min pre-dose and at 5 min, 10 min, 25 min and 50 min post-dose
Population: Treated set (observed cases)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | Tio+Olo 5/5μg | Tiotropium 5μg + Olodaterol 5μg
Number analyzed (Participants) | 52 | 52 | 52
ms
  5 min | -0.3 (1.5) | -0.2 (1.8) | -0.0 (1.6)
  10 min | -0.3 (1.6) | 0.1 (1.6) | 0.1 (1.6)
  25 min | -0.3 (1.4) | 0.1 (1.6) | 0.0 (1.4)
  50 min | -0.4 (1.7) | 0.2 (1.7) | 0.2 (1.6)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) occurring up to the minimum of 21 days after drug stop date or the start of the next treatment period were considered on treatment; Up to 64 days.
Groups:
- Tio+Olo FDC: Single test dose of oral inhalation of Tio+Olo FDC(fixed dose combination) (5/5 μg) inhalation solution as fixed dose inhalation solution (Tio+Olo FDC) 2.5 μg each per actuation via RESPIMAT inhaler.
  2 inhalations a.m. dosing.
- Tiotropium and Olodaterol FC: Single test dose of oral inhalation of tiotropium (5 μg) and olodaterol (5 μg) free combination FC (Tio/Olo free combination)
  Olodaterol: 5 μg (2.5 μg per actuation)
  Tiotropium: 5 μg (2.5 μg per actuation)
  2 inhalations a.m. dosing.
Arm/Group | Placebo | Tio+Olo FDC | Tiotropium and Olodaterol FC
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/52 | 2/52
Other Adverse Events (participants affected / at risk) | 3/53 | 1/52 | 2/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=53) | Tio+Olo FDC (N=52) | Tiotropium and Olodaterol FC (N=52)
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=53) | Tio+Olo FDC (N=52) | Tiotropium and Olodaterol FC (N=52)
Nasopharyngitis (Infections and infestations) | 3 | 1 | 2

LIMITATIONS AND CAVEATS:
Additional secondary endpoints were listed in the original protocol. Those endpoints are of exploratory nature only and were not considered relevant for trial conclusions. For more information see tab "Full Text Review", section "More Information".

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.